CLINICAL TRIAL: NCT00195910
Title: Safety and Efficacy of Hydromorphone as an Analgesic Alternative to Morphine in Acute, Severe Pain: A Randomized Clinical Trial
Brief Title: Safety and Efficacy Study of Hydromorphone and Morphine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC-04-08-225
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Acute; Pain; Emergency Department; Morphine; Hydromorphone; Dilaudid; oligoanalgesia
MeSH Terms: conditions — Pain; Emergencies | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Morphine (Active Comparator): single dose of intravenous (IV) morphine, 0.1 mg/kg
  intervention: 0.1 mg/kg IV morphine
  Interventions: Drug: Morphine
- Hydromorphone (Experimental): single dose of intravenous (IV) hydromorphone, 0.015 mg/kg
  intervention: 0.015 mg/kg IV hydromorphone
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Morphine — 0.1 mg/kg IV morphine
  Arms: Morphine
Drug: Hydromorphone — 0.015 mg/kg IV hydromorphone
  Other Names: Dilaudid
  Arms: Hydromorphone

SUMMARY:
To compare a standard weight-based dose of intravenous (IV) hydromorphone (Dilaudid) to a standard weight-based dose of IV morphine in adults presenting to the Emergency Department (ED) with acute severe pain.

DETAILED DESCRIPTION:
There is widespread agreement that pain is under-treated in the Emergency Department (ED). The current recommended treatment of acute pain in the ED setting is administration of an initial bolus of morphine followed by titration until adequate analgesia is achieved. Several studies have shown that even 0.1 mg/kg IV morphine (7-10 mg administered to the average 70-100 kg patient) inadequately treats many patients' acute pain. In spite of this, it has been observed that many emergency physicians and nurses are hesitant to give 7-10 mg of morphine as an initial IV dose. In contrast, it has been observed that these same healthcare providers were not similarly reluctant to administer a roughly equianalgesic dose of hydromorphone (1-1.5 mg), perhaps because the more potent hydromorphone is given in much smaller milligram quantities than morphine, thus providing the illusion of substantially less opioid administered to the patient. Having repeatedly observed this phenomenon, it is reasonable that if a smaller milligram dose of hydromorphone were shown to provide an efficacy, safety, and side-effect profile comparable or superior to a larger milligram dose of morphine, it would provide evidence supporting use of hydromorphone as an alternative first line opioid in the treatment of acute pain presenting to the ED. As a practical corollary to this, it is reasoned further that the increased willingness of healthcare providers to use hydromorphone might contribute to reducing one component of the multifaceted problem of oligoanalgesia in the ED.

ELIGIBILITY:
Inclusion Criteria:

* adults between the ages of 21 and 65 who presented to the ED with acute pain (defined as pain less than 7 days in duration) (23) of sufficient severity in the judgment of the ED attending to warrant use of IV opioids.

Exclusion Criteria:

* previous allergy to morphine or hydromorphone
* systolic blood pressure less than 90 mmHg
* alcohol intoxication as judged by the attending physician
* use of other opioids within the past 7 days
* use of an Monoamine Oxidase (MAO) inhibitor
* chronic pain syndromes (such as sickle cell disease or fibromyalgia)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity from baseline to 30 minutes after medications were infused. | baseline to 30 minutes after medication infused
  Pain intensity is measured by the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Pain intensity 5 minutes after medication is given | 5 minutes after medication is given
  Pain intensity is measured by the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Pain intensity 30 minutes after medication is given | 30 minutes after medication is given
  Pain intensity is measured by the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Pain intensity 2 hours after medication is given | 2 hours after medication is given
  Pain intensity is measured by the numerical rating scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Number of participants experiencing vomiting between baseline to 5 minutes after medication is given | baseline to 5 minutes after medication is given
  Number of participants who experienced vomiting and required medication between baseline and 5 minutes after medication was infused
Number of participants experiencing vomiting between 6 minutes after medication is given to 30 minutes after medication is given | 6 minutes after medication is given to 30 minutes after medication is given
  Number of participants who experienced vomiting and required medication between 6 minutes after medication was infused and 30 minutes after medication was infused
Number of participants experiencing vomiting between 31 minutes after medication is given to 120 minutes after medication is given | 31 minutes after medication is given to 120 minutes after medication is given
  Number of participants who experienced vomiting and required medication between 31 minutes after medication was infused and 120 minutes after medication was infused
Number of participants who received additional pain medication between baseline and 5 minutes after medication was infused | baseline to 5 minutes after medication was infused
  Number of participants for whom the administered pain medication was not sufficient, leading to the patient receiving additional pain medication between baseline and 5 minutes after medication was infused
Number of participants who received additional pain medication between 6 and 30 minutes after medication was infused | 6 minutes to 30 minutes after medication was infused
  Number of patients for whom the administered pain medication was not sufficient, leading to the patient receiving additional pain medication between 6 and 30 minutes after the medication was infused
Number of participants who received additional pain medication between 31 and 120 minutes after medication was infused | 31 minutes to 120 minutes after medication was infused
  Number of patients for whom the administered pain medication was not sufficient, leading to the patient receiving additional pain medication between 31 and 120 minutes after medication was infused

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Chang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States